CLINICAL TRIAL: NCT05197751
Title: Phase 1 Randomized, Dose-finding Study to Evaluate the Safety, Tolerability and Immunogenicity of a Novel Malaria Vaccine, MSP3-CRM-Vac4All/ Alhydrogel®, in Healthy Adults
Brief Title: MSP3-CRM-Vac4All/ Alhydrogel® Malaria Vaccine
Acronym: MSP3CRMV4All
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vac4All (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V4ALL/MSP3/008
Record Dates: First submitted 2021-11-24; First posted 2022-01-19 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Aluminum Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 µg dose cohort (Experimental): 3 µg MSP3-CRM-Vac4All/Alhydrogel®
  Interventions: Biological: MSP3-CRM-Vac4All/ Alhydrogel®
- 10 µg dose cohort (Experimental): 10 µg MSP3-CRM-Vac4All/Alhydrogel®
  Interventions: Biological: MSP3-CRM-Vac4All/ Alhydrogel®
- 30 µg dose cohort (Experimental): 30 µg MSP3-CRM-Vac4All/Alhydrogel®
  Interventions: Biological: MSP3-CRM-Vac4All/ Alhydrogel®

INTERVENTIONS:
Biological: MSP3-CRM-Vac4All/ Alhydrogel® — The Investigational Medicinal Product (IMP) or in short Investigational Product (IP) is the MSP3-CRM-Vac4All/ Alhydrogel® vaccine

SUMMARY:
First-in-Human, Randomised, Dose-Finding Single Center Study to evaluate three dose levels of a novel malaria vaccine, MSP3-CRM-Vac4All/ Alhydrogel® : 3 µg, 10 µg and 30 µg

DETAILED DESCRIPTION:
A total of 42 healthy male and female participants aged 18 to 55 years will be enrolled and randomized into one of three cohorts. Three dose levels of a novel malaria vaccine, MSP3-CRM-Vac4All/ Alhydrogel®, will be evaluated: 3 µg, 10 µg and 30 µg total MSP3-CRM197 conjugate protein (corresponding to 1, 3, 10 µg MSP3 protein) administered as a primary series of three intramuscular (IM) injections, given on day 1, day 28, and day 56.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-55 years old
* In general good health by medical history, physical examination and laboratory investigation
* Resident in the study area for the duration of the study with mobile phone access (personal or family) during the first 4 months of trial participation.
* Negative pregnancy test and the use of effective contraception during the whole study period if deemed appropriate.
* Willingness to undergo an HIV test.
* Signed informed consent following demonstration of proper understanding of the meaning and procedures of the First-in-Human Phase I trial.

Exclusion Criteria:

* Any history of documented malaria over the last 3 years.
* Born and lived till adolescence (up to 15 years) in rural high transmission malaria endemic area
* Any plans to travel and stay in malaria endemic areas during the study period for more than one week.
* Positivity by Elisa at screening on either MSP3-C terminal antigen, or AMA1, or LSA3-R, or EBA 175 (positivity defined as optical density (OD) as high or higher than lower threshold of positivity post 1st generation MSP3 in Doneguebougou)
* Use of any investigational drug or vaccine other than the study vaccine within 30 days before the first dose up to 30 days after third and last dose of vaccination.
* Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior recruitment or planned administration during study period (for corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* Planned administration of any other vaccine not foreseen by the study protocol within 30 days before the first dose up to 30 days after third and last dose of vaccination. Some biologicals may be administered as emergency measure during the trial, such as tetanus toxoid or serum, rabies vaccine and immunoglobulins
* Suspected or known hypersensitivity or allergic reactions to any of the vaccine components or to previous vaccine.
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis.
* Symptoms, physical signs and laboratory values suggestive of past or current history of significant neurological, cardiovascular, pulmonary, hepatic, rheumatic, autoimmune, hematological, metabolic, renal, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers
* Seropositive for HIV at screening
* Presence of chronic illness that, in the judgment of the investigator, would interfere with the study outcomes or pose a threat to the participant's health.
* History of surgical splenectomy.
* Moderate or severe malnutrition at screening based on appropriate Body Mass Index (BMI) thresholds (to be defined by site).
* Cannot be followed for any social, psychological or geographical reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-05-09 (Estimated)

PRIMARY OUTCOMES:
To measure the frequency and grade of each solicited local and systemic reactions during the 7 days following each vaccination of MSP3-CRM-Vac4All/ Alhydrogel® for each dose levels (3 µg, 10 µg and 30 µg), administered on Day 1, 28 and 56 | Over 7 days following vaccination
  Frequency and grade of each solicited local and systemic reactions during the 7 days following each vaccination, for each treatment group.
To measure the frequency and grade of any unsolicited AEs during the 28 days following each vaccination of MSP3-CRM-Vac4All/ Alhydrogel® for each dose levels (3 µg, 10 µg and 30 µg), administered on Day 1, 28 and 56 | Over 28 days following vaccination
  Frequency and grade of any unsolicited AEs during the 28 days following each vaccination, for each treatment group.
To measure the frequency of Serious Adverse Events (AEs) following the first dose of the vaccine until the last follow-up visit. | Over 12 month following first vaccination
  Frequency of Serious Adverse Events (AEs) observed from the first dose of the vaccine until the last follow-up visit.
To measure the number of subjects with Adverse Events (AEs) during the 28 days following each vaccination, for each dose levels (3 µg, 10 µg and 30 µg), administered on Day 1, 28 and 56 | Over 28 days following vaccination
  Number of subjects with Adverse Events (AEs) during the 28 days following each vaccination, for each treatment group.

SECONDARY OUTCOMES:
To measure the frequency and grade of each solicited systemic and local reaction during the 7 days following each vaccination, for the combined active vaccination group | 7 days following vaccination
  Frequency and grade of solicited systemic and local reaction during the 7 days following each vaccination, for the combined active vaccination group.
To measure the frequency and grade of each unsolicited systemic and local reaction during the 28 days for the combined active vaccination group of each dose levels (3 µg, 10 µg and 30 µg), administered on Day 1, 28 and 56 | 28 days following vaccination
  Frequency and grade of unsolicited systemic and local reaction during the 28 days following each vaccination, for the combined active vaccination group.
To measure the number of subjects with Adverse Events during the 28 days each vaccination, for the combined active vaccination group. | 28 days after vaccination
  the number of subjects with Adverse Events during the 28 days each vaccination, for the combined active vaccination group.
To measure the seroresponse rates (defined as the proportion with 2, 3, and 4-fold rise in titre of anti-MSP3 antibodies) determined 28 days after each vaccination as compared to baseline (Day 1), by treatment group. | 28 days after vaccination
  Seroresponse rates (defined as the proportion with 2, 3, and 4-fold rise in titre of anti-MSP3 antibodies) determined 28 days after each vaccination as compared to baseline (Day 1), by treatment group.
To measure the Geometric mean titres (GMT) of anti-MSP3 antibodies 28 days after each vaccination, by treatment group (total IgG and IgG sub classes).observed during the 28 days following each vaccination, for the combined active vaccination group. | 28 days after each vaccination
  Geometric mean titres (GMT) of anti-MSP3 antibodies 28 days after each vaccination, by treatment group (total IgG and IgG sub classes).
To measure Geometric mean fold increase (GMFI) of anti-MSP3 antibodies determined 28 days after each vaccination as compared to baseline (total IgG and IgG sub classes). | 28 days after each vaccination
  Geometric mean fold increase (GMFI) of anti-MSP3 antibodies determined 28 days after each vaccination as compared to baseline (total IgG and IgG sub classes).
To measure the Proportion of participants with seroresponse across all time points | one month, 3 months, 6 months and 12 months after first vaccination
  Proportion of participants with seroresponse across all time points
To measure the Seroresponse rates, GMTs and GMFI of anti-MSP3 antibodies 3, 6 and 12 months after first vaccination (total IgG and IgG sub classes). | 3, 6 and 12 month after first vaccination
  Seroresponse rates, GMTs and GMFI of anti-MSP3 antibodies 3, 6 and 12 months after first vaccination (total IgG and IgG sub classes).
To measureIgG ability to recognize the native protein on merozoite by using Western Blot (WB) and IFAT methods | one month after each vaccination and 3 months, 6 months and 12 months after first vaccination
  IgG ability to recognize the native protein on merozoite by using Western Blot (WB) and IFAT methods

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou Thera, MD, Study Director — MRTC, University of Sciences Techniques and Technologies of Bamako, Mali
Locations (1):
- Malaria Research and Training Center (MRTC), University of Sciences Techniques and Technologies of Bamako, Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No